CLINICAL TRIAL: NCT05064397
Title: Interventional, Open-label, Fixed-dose Multiple Administration Study to Evaluate Long-term Treatment With Eptinezumab in Patients With Chronic Cluster Headache
Brief Title: A 1-year Trial to Inform About Long-term Exposure to Eptinezumab in Participants With Chronic Cluster Headache (cCH)
Acronym: CHRONICLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19385A
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Chronic Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — eptinezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eptinezumab (Experimental): Participants will receive 4 intravenous (IV) infusions with eptinezumab at Baseline (Day 0) and at the end of Weeks 12, 24, and 36.
  Interventions: Drug: Eptinezumab

INTERVENTIONS:
Drug: Eptinezumab — Eptinezumab will be administered per schedule specified in the arm description.
  Other Names: Vyepti

SUMMARY:
The main goal of this trial is to inform about long-term safety and tolerability of eptinezumab in participants with chronic cluster headache.

DETAILED DESCRIPTION:
The participants who take part in this trial will be asked to stay in the trial for about a year. The participants will be asked to visit the trial site 7 times during the trial. In between trial site visits, they will have scheduled phone calls with the trial site staff. They will also be asked to keep track of their cluster headaches at home with a headache diary.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a diagnosis of cCH as defined by International Headache Society (IHS) International Classification of Headache Disorders third edition (ICHD-3) classification with a history of cCH of at least 12 months prior to the Screening Visit.
* The participant has a medical history of onset of cluster headache at ≤50 years of age.
* The participant has an adequately documented record of previous abortive, transitional and preventive medication use for cCH, for at least 12 months prior to the Screening Visit.
* The participant is able to distinguish cluster headache attacks from other headaches (such as tension-type headaches, migraine).

Exclusion Criteria:

* The participant has experienced failure on a previous treatment targeting the calcitonin gene-related peptide (CGRP) pathway (anti-CGRP monoclonal antibodies [mAbs] and gepants).
* The participant has confounding and clinically significant pain syndromes (for example, fibromyalgia, complex regional pain syndrome).
* The participant has a history or diagnosis of chronic tension-type headache, hypnic headache, hemicrania continua, new daily persistent headache, chronic migraine or unusual migraine subtypes such as hemiplegic migraine (sporadic and familial), recurrent painful ophthalmoplegic neuropathy, migraine with neurological accompaniments that are not typical of migraine aura (diplopia, altered consciousness, or longer than 1 hour).
* Participants with a lifetime history of psychosis, bipolar mania, or dementia. Participants with other psychiatric conditions whose symptoms are not controlled or who have not been adequately treated for a minimum of 6 months prior to Screening Visit.
* The participant has attempted suicide or is, at Screening Visit, at significant risk of suicide.
* The participant has a history of clinically significant cardiovascular disease, including uncontrolled hypertension, vascular ischaemia or thromboembolic events (for example, cerebrovascular accident, deep vein thrombosis, or pulmonary embolism).

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (31):
- United States (5):
  - New England Institute for Neurology and Headache, Stamford, Connecticut
  - Michigan Headache and Neurological Institute, Ann Arbor, Michigan
  - Dent Neurologic Institute - Amherst, Amherst, New York
  - Cleveland Clinic - Neurological Institute, Cleveland, Ohio
  - Thomas Jefferson University Hospital - Center City Campus, Philadelphia, Pennsylvania
- Denmark (2):
  - Rigshospitalet Glostrup, Glostrup Municipality, Capital Region
  - Hospitalsenhed Midt og Regionshospitalet Viborg, Viborg, Central Jutland
- Finland (2):
  - Terveystalo Ruoholahti, Helsinki, Southern Finland
  - Terveystalo Turku Pulssi, Turku, Western Finland
- France (6):
  - Hôpital Cimiez, Nice, Côte-d'Or
  - Hôpital Roger Salengro, Lille, Nord
  - Hôpital de la Timone, Marseille, Provence-Alpes-Côte d'Azur Region
  - Hôpital Pierre Wertheimer, Bron, Rhône
  - Centre Hospitalier Universitaire de Saint-Étienne, Saint-Priest-en-Jarez, Rhône
  - Hôpital Lariboisière, Paris, Île-de-France Region
- Germany (2):
  - Kopfschmerzzentrum Frankfurt, Frankfurt am Main, Hesse
  - Charité Campus Mitte, Berlin
- Italy (5):
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Fondazione Istituto Neurologico Car..., Milan, Milan
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - San Raffaele Pisana, Rome, Roma
  - IRCCS Istituto Delle Scienze Neurologiche di Bologna, Bologna
  - Fondazione Mondino - Istituto Neurologico Nazionale a Carattere Scientifico IRCCS, Pavia
  - Ospedale Molinette - Clinica Neurologica II - Centro Cefalee, Turin
- Netherlands (2):
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Brain Research Center - Amsterdam, Amsterdam, North Holland
- Spain (5):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
- United Kingdom (2):
  - The Walton Centre NHS Foundation Trust, Liverpool, England
  - King's College Hospital NHS Foundation Trust, London, England

REFERENCES:
- [Derived] Tassorelli C, Jensen RH, Goadsby PJ, Charles AC, Tepper SJ, Snoer AH, Josiassen MK, Linander CB, Ettrup A, Sperling B, Boneva N. Long-term safety, tolerability, and efficacy of eptinezumab in chronic cluster headache (CHRONICLE): an open-label safety trial. Lancet Neurol. 2025 May;24(5):429-440. doi: 10.1016/S1474-4422(25)00065-1. PMID 40252664

RESULTS

PARTICIPANT FLOW:
Groups:
- Eptinezumab: Participants received 4 intravenous (IV) infusions of 400 milligrams (mg) eptinezumab at Baseline (Day 0) and at the end of Weeks 12, 24, and 36.
Period: Overall Study
Arm/Group | Eptinezumab
Started | 131
Received at Least 1 Dose of Study Drug | 131
Completed | 108
Not Completed | 23
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 12
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1
Not completed — Other reasons | 3

BASELINE CHARACTERISTICS:
Population: The all-participants-treated set (APTS) included all participants who received infusion with eptinezumab.
Groups:
- Eptinezumab: Participants received 4 IV infusions of 400 mg eptinezumab at Baseline (Day 0) and at the end of Weeks 12, 24, and 36.
Arm/Group | Eptinezumab
Number analyzed (Participants) | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 76
  More than one race | 4
  Unknown or Not Reported | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs)
Description: A treatment-emergent AE was defined as any on-treatment untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A summary of non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: From the day of first dose of study drug (Baseline [Week 0]) up to Week 56
Population: The APTS included all participants who received infusion with eptinezumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab
Number analyzed (Participants) | 131
Participants | 106

2. Secondary Outcome: Conversion From Chronic Cluster Headache (cCH) to Episodic Cluster Headache (eCH): Number of Participants With No Cluster Headache (CH) Attacks for ≥3 Consecutive Months (≥12 Consecutive Weeks)
Description: Participants counted as converting from cCH to eCH if they had no CH attacks for at least 3 months.
Time Frame: Week 1 to Week 48
Population: The Full Analysis Set (FAS) included all participants in the APTS who had a valid assessment of the baseline number of weekly attacks and a post-baseline assessment of the number of weekly attacks.
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab
Number analyzed (Participants) | 131
Participants | 7

3. Secondary Outcome: Change From Baseline in Weekly Number of Times an Abortive Therapy (Oxygen and/or Triptans) Was Used
Description: Abortive therapy was defined as oxygen and/or triptans, where it counted as 2 times if oxygen and triptans were used for the same attack.
Time Frame: Baseline (Week 0), Weeks 1, 2, 3, 4, 13, 14, 15, 16, 25, 26, 27, 28, 37, 38, 39, 40
Population: The FAS included all participants in the APTS who had a valid assessment of the baseline number of weekly attacks and a post-baseline assessment of the number of weekly attacks. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure, and "Number analyzed" is the number of participants evaluable at each specified time point.
Measure: Least Squares Mean (Standard Error); unit: Abortive therapy use per week
Arm/Group | Eptinezumab
Number analyzed (Participants) | 127
Abortive therapy use per week
  Week 1 | -3.63 (0.53)
  Week 2: number analyzed (Participants) | 123
  Week 2 | -4.24 (0.70)
  Week 3: number analyzed (Participants) | 117
  Week 3 | -4.90 (0.76)
  Week 4: number analyzed (Participants) | 110
  Week 4 | -4.99 (0.94)
  Week 13: number analyzed (Participants) | 93
  Week 13 | -7.22 (0.84)
  Week 14: number analyzed (Participants) | 101
  Week 14 | -6.83 (0.85)
  Week 15: number analyzed (Participants) | 95
  Week 15 | -6.06 (0.84)
  Week 16: number analyzed (Participants) | 89
  Week 16 | -6.42 (0.96)
  Week 25: number analyzed (Participants) | 96
  Week 25 | -6.18 (0.99)
  Week 26: number analyzed (Participants) | 93
  Week 26 | -6.56 (0.86)
  Week 27: number analyzed (Participants) | 89
  Week 27 | -7.56 (0.82)
  Week 28: number analyzed (Participants) | 81
  Week 28 | -7.12 (0.83)
  Week 37: number analyzed (Participants) | 87
  Week 37 | -6.55 (0.98)
  Week 38: number analyzed (Participants) | 87
  Week 38 | -6.97 (0.84)
  Week 39: number analyzed (Participants) | 77
  Week 39 | -6.71 (1.04)
  Week 40: number analyzed (Participants) | 70
  Week 40 | -7.09 (0.84)

4. Secondary Outcome: Change From Baseline in Weekly Number of Times An Abortive Therapy (Oxygen) Was Used
Time Frame: Baseline (Week 0), Weeks 1, 2, 3, 4, 13, 14, 15, 16, 25, 26, 27, 28, 37, 38, 39, 40
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Oxygen use per week
Arm/Group | Eptinezumab
Number analyzed (Participants) | 127
Oxygen use per week
  Week 1 | -1.72 (0.33)
  Week 2: number analyzed (Participants) | 123
  Week 2 | -2.43 (0.40)
  Week 3: number analyzed (Participants) | 117
  Week 3 | -3.17 (0.48)
  Week 4: number analyzed (Participants) | 110
  Week 4 | -3.23 (0.59)
  Week 13: number analyzed (Participants) | 93
  Week 13 | -3.97 (0.57)
  Week 14: number analyzed (Participants) | 101
  Week 14 | -3.93 (0.56)
  Week 15: number analyzed (Participants) | 95
  Week 15 | -3.09 (0.53)
  Week 16: number analyzed (Participants) | 89
  Week 16 | -3.78 (0.61)
  Week 25: number analyzed (Participants) | 96
  Week 25 | -3.56 (0.67)
  Week 26: number analyzed (Participants) | 93
  Week 26 | -3.75 (0.58)
  Week 27: number analyzed (Participants) | 89
  Week 27 | -4.06 (0.52)
  Week 28: number analyzed (Participants) | 81
  Week 28 | -4.02 (0.54)
  Week 37: number analyzed (Participants) | 87
  Week 37 | -3.60 (0.64)
  Week 38: number analyzed (Participants) | 87
  Week 38 | -3.74 (0.52)
  Week 39: number analyzed (Participants) | 77
  Week 39 | -3.99 (0.66)
  Week 40: number analyzed (Participants) | 70
  Week 40 | -3.82 (0.55)

5. Secondary Outcome: Change From Baseline in Weekly Number of Times An Abortive Therapy (Triptans) Were Used
Time Frame: Baseline (Week 0), Weeks 1, 2, 3, 4, 13, 14, 15, 16, 25, 26, 27, 28, 37, 38, 39, 40
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Triptans use per week
Arm/Group | Eptinezumab
Number analyzed (Participants) | 127
Triptans use per week
  Week 1 | -1.75 (0.33)
  Week 2: number analyzed (Participants) | 123
  Week 2 | -1.73 (0.42)
  Week 3: number analyzed (Participants) | 117
  Week 3 | -1.74 (0.44)
  Week 4: number analyzed (Participants) | 110
  Week 4 | -1.90 (0.45)
  Week 13: number analyzed (Participants) | 93
  Week 13 | -2.94 (0.46)
  Week 14: number analyzed (Participants) | 101
  Week 14 | -2.78 (0.50)
  Week 15: number analyzed (Participants) | 95
  Week 15 | -2.81 (0.49)
  Week 16: number analyzed (Participants) | 89
  Week 16 | -2.50 (0.51)
  Week 25: number analyzed (Participants) | 96
  Week 25 | -2.05 (0.52)
  Week 26: number analyzed (Participants) | 93
  Week 26 | -2.48 (0.48)
  Week 27: number analyzed (Participants) | 89
  Week 27 | -3.06 (0.45)
  Week 28: number analyzed (Participants) | 81
  Week 28 | -2.86 (0.46)
  Week 37: number analyzed (Participants) | 87
  Week 37 | -2.55 (0.50)
  Week 38: number analyzed (Participants) | 87
  Week 38 | -2.54 (0.49)
  Week 39: number analyzed (Participants) | 77
  Week 39 | -2.52 (0.58)
  Week 40: number analyzed (Participants) | 70
  Week 40 | -2.95 (0.54)

6. Secondary Outcome: Change From Baseline in the Average Number of Weekly Attacks
Description: The participant completed a CH eDiary, daily, and record for each day/week whether he/she had any CH attacks.
Time Frame: Baseline (Week 0), Weeks 1, 2, 3, 4, 13, 14, 15, 16, 25, 26, 27, 28, 37, 38, 39, 40
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Attacks per week
Arm/Group | Eptinezumab
Number analyzed (Participants) | 127
Attacks per week
  Week 1 | -3.00 (0.54)
  Week 2: number analyzed (Participants) | 123
  Week 2 | -3.92 (0.79)
  Week 3: number analyzed (Participants) | 117
  Week 3 | -4.51 (0.93)
  Week 4: number analyzed (Participants) | 110
  Week 4 | -4.98 (1.18)
  Week 13: number analyzed (Participants) | 93
  Week 13 | -6.18 (1.20)
  Week 14: number analyzed (Participants) | 101
  Week 14 | -6.31 (1.15)
  Week 15: number analyzed (Participants) | 95
  Week 15 | -5.81 (1.08)
  Week 16: number analyzed (Participants) | 89
  Week 16 | -6.63 (1.24)
  Week 25: number analyzed (Participants) | 96
  Week 25 | -5.56 (1.26)
  Week 26: number analyzed (Participants) | 93
  Week 26 | -5.95 (1.27)
  Week 27: number analyzed (Participants) | 89
  Week 27 | -7.09 (1.22)
  Week 28: number analyzed (Participants) | 81
  Week 28 | -6.51 (1.31)
  Week 37: number analyzed (Participants) | 87
  Week 37 | -6.25 (1.27)
  Week 38: number analyzed (Participants) | 87
  Week 38 | -6.57 (1.14)
  Week 39: number analyzed (Participants) | 77
  Week 39 | -5.99 (1.23)
  Week 40: number analyzed (Participants) | 70
  Week 40 | -6.39 (1.15)

7. Secondary Outcome: Change From Baseline in the Number of Weekly Attacks
Description: The average of the estimated change from baseline in the number of weekly attacks across the first 4 weeks after the infusion is shown.
Time Frame: Baseline (Week 0), Weeks 1-4
Population: The FAS included all participants in the APTS who had a valid assessment of the baseline number of weekly attacks and a post-baseline assessment of the number of weekly attacks. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Attacks per week
Arm/Group | Eptinezumab
Number analyzed (Participants) | 127
Attacks per week | -4.11 (0.79)

8. Secondary Outcome: Change From Baseline in the Number of Weekly Attacks
Description: The average of the estimated change from baseline in the number of weekly attacks across the first 2 weeks after the infusion is shown.
Time Frame: Baseline (Week 0), Weeks 1-2
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Attacks per week
Arm/Group | Eptinezumab
Number analyzed (Participants) | 127
Attacks per week | -3.46 (0.61)

9. Secondary Outcome: Change From Baseline in the Number of Monthly Attacks
Description: The average of the estimated change from baseline in the number of monthly attacks across the first 12 months after the infusion is shown.
Time Frame: Baseline (Week 0), Months 1-12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Attacks per month
Arm/Group | Eptinezumab
Number analyzed (Participants) | 129
Attacks per month | -22.65 (4.39)

10. Secondary Outcome: Change From Baseline in the Average Attack Related Daily Pain (Including Days With no Attacks), as Assessed Using the 5-point Self-rating Pain Severity Scale
Description: The severity of pain for each attack was rated on an ordinal scale that ranged from 0 to 4 with higher scores indicating more headache pain (headache pain ratings: 0 = none/barely any pain; 1 = mild; 2 = moderate; 3 = severe; 4 = excruciating).
Time Frame: Baseline (Week 0), Weeks 1, 2, 3, 4, 13, 14, 15, 16, 25, 26, 27, 28, 37, 38, 39, 40
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Eptinezumab
Number analyzed (Participants) | 127
score on a scale
  Week 1 | -0.47 (0.06)
  Week 2: number analyzed (Participants) | 123
  Week 2 | -0.51 (0.07)
  Week 3: number analyzed (Participants) | 117
  Week 3 | -0.58 (0.07)
  Week 4: number analyzed (Participants) | 110
  Week 4 | -0.59 (0.08)
  Week 13: number analyzed (Participants) | 93
  Week 13 | -0.78 (0.09)
  Week 14: number analyzed (Participants) | 101
  Week 14 | -0.75 (0.09)
  Week 15: number analyzed (Participants) | 95
  Week 15 | -0.82 (0.08)
  Week 16: number analyzed (Participants) | 89
  Week 16 | -0.90 (0.09)
  Week 25: number analyzed (Participants) | 96
  Week 25 | -0.80 (0.09)
  Week 26: number analyzed (Participants) | 93
  Week 26 | -0.79 (0.09)
  Week 27: number analyzed (Participants) | 89
  Week 27 | -0.88 (0.09)
  Week 28: number analyzed (Participants) | 81
  Week 28 | -0.84 (0.09)
  Week 37: number analyzed (Participants) | 87
  Week 37 | -0.77 (0.09)
  Week 38: number analyzed (Participants) | 87
  Week 38 | -0.79 (0.10)
  Week 39: number analyzed (Participants) | 77
  Week 39 | -0.70 (0.10)
  Week 40: number analyzed (Participants) | 70
  Week 40 | -0.79 (0.10)

11. Secondary Outcome: Response: Number of Participants With ≥30% Reduction From Baseline in Number of Weekly Attacks
Time Frame: Baseline (Week 0), Weeks 1, 2, 3, 4, 13, 14, 15, 16, 25, 26, 27, 28, 37, 38, 39, 40
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab
Number analyzed (Participants) | 127
Participants
  Week 1 | 49
  Week 2: number analyzed (Participants) | 123
  Week 2 | 52
  Week 3: number analyzed (Participants) | 117
  Week 3 | 55
  Week 4: number analyzed (Participants) | 110
  Week 4 | 55
  Week 13: number analyzed (Participants) | 93
  Week 13 | 54
  Week 14: number analyzed (Participants) | 101
  Week 14 | 63
  Week 15: number analyzed (Participants) | 95
  Week 15 | 58
  Week 16: number analyzed (Participants) | 89
  Week 16 | 62
  Week 25: number analyzed (Participants) | 96
  Week 25 | 60
  Week 26: number analyzed (Participants) | 93
  Week 26 | 60
  Week 27: number analyzed (Participants) | 89
  Week 27 | 62
  Week 28: number analyzed (Participants) | 81
  Week 28 | 48
  Week 37: number analyzed (Participants) | 87
  Week 37 | 57
  Week 38: number analyzed (Participants) | 87
  Week 38 | 51
  Week 39: number analyzed (Participants) | 77
  Week 39 | 43
  Week 40: number analyzed (Participants) | 70
  Week 40 | 44

12. Secondary Outcome: Response: Number of Participants With ≥50% Reduction From Baseline in Number of Weekly Attacks
Time Frame: Baseline (Week 0), Weeks 1, 2, 3, 4, 13, 14, 15, 16, 25, 26, 27, 28, 37, 38, 39, 40
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab
Number analyzed (Participants) | 127
Participants
  Week 1 | 30
  Week 2: number analyzed (Participants) | 123
  Week 2 | 36
  Week 3: number analyzed (Participants) | 117
  Week 3 | 42
  Week 4: number analyzed (Participants) | 110
  Week 4 | 40
  Week 13: number analyzed (Participants) | 93
  Week 13 | 35
  Week 14: number analyzed (Participants) | 101
  Week 14 | 45
  Week 15: number analyzed (Participants) | 95
  Week 15 | 43
  Week 16: number analyzed (Participants) | 89
  Week 16 | 48
  Week 25: number analyzed (Participants) | 96
  Week 25 | 43
  Week 26: number analyzed (Participants) | 93
  Week 26 | 45
  Week 27: number analyzed (Participants) | 89
  Week 27 | 45
  Week 28: number analyzed (Participants) | 81
  Week 28 | 39
  Week 37: number analyzed (Participants) | 87
  Week 37 | 40
  Week 38: number analyzed (Participants) | 87
  Week 38 | 41
  Week 39: number analyzed (Participants) | 77
  Week 39 | 34
  Week 40: number analyzed (Participants) | 70
  Week 40 | 38

13. Secondary Outcome: Response: Number of Participants With ≥75% Reduction From Baseline in Number of Weekly Attacks
Time Frame: Baseline (Week 0), Weeks 1, 2, 3, 4, 13, 14, 15, 16, 25, 26, 27, 28, 37, 38, 39, 40
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab
Number analyzed (Participants) | 127
Participants
  Week 1 | 11
  Week 2: number analyzed (Participants) | 123
  Week 2 | 13
  Week 3: number analyzed (Participants) | 117
  Week 3 | 21
  Week 4: number analyzed (Participants) | 110
  Week 4 | 20
  Week 13: number analyzed (Participants) | 93
  Week 13 | 23
  Week 14: number analyzed (Participants) | 101
  Week 14 | 25
  Week 15: number analyzed (Participants) | 95
  Week 15 | 23
  Week 16: number analyzed (Participants) | 89
  Week 16 | 29
  Week 25: number analyzed (Participants) | 96
  Week 25 | 29
  Week 26: number analyzed (Participants) | 93
  Week 26 | 24
  Week 27: number analyzed (Participants) | 89
  Week 27 | 28
  Week 28: number analyzed (Participants) | 81
  Week 28 | 24
  Week 37: number analyzed (Participants) | 87
  Week 37 | 27
  Week 38: number analyzed (Participants) | 87
  Week 38 | 28
  Week 39: number analyzed (Participants) | 77
  Week 39 | 21
  Week 40: number analyzed (Participants) | 70
  Week 40 | 25

14. Secondary Outcome: cCH Remission: Number of Participants With No Cluster Headache Attacks For ≥1 Month (>=4 Consecutive Weeks)
Description: Participants counted as being in remission if they had no cluster headache attacks for at least 1 month.
Time Frame: Week 1 to Week 48
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab
Number analyzed (Participants) | 131
Participants | 19

15. Secondary Outcome: cCH Remission: Number of Participants With No Cluster Headache Attacks For ≥1 Month (>=4 Consecutive Weeks Between the First and Second Infusion)
Time Frame: Week 1 to Week 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab
Number analyzed (Participants) | 129
Participants | 8

16. Secondary Outcome: cCH Remission: Number of Participants With No Cluster Headache Attacks For ≥1 Month (>=4 Consecutive Weeks Between the Second and Third Infusion)
Time Frame: Week 13 to Week 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab
Number analyzed (Participants) | 119
Participants | 10

17. Secondary Outcome: cCH Remission: Number of Participants With No Cluster Headache Attacks For ≥1 Month (>=4 Consecutive Weeks Between the Third and Fourth Infusion)
Time Frame: Week 25 to Week 36
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab
Number analyzed (Participants) | 111
Participants | 9

18. Secondary Outcome: cCH Remission: Number of Participants With No Cluster Headache Attacks For ≥1 Month (>=4 Consecutive Weeks Within the First 12 Weeks After the Fourth Infusion)
Time Frame: Week 37 to Week 48
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab
Number analyzed (Participants) | 104
Participants | 10

19. Secondary Outcome: Number of Participants Who Received a Transitional Therapy During the Treatment Period
Description: Transitional treatments were defined as greater occipital nerve (GON) block or oral steroids.
Time Frame: Week 1 to Week 48
Population: The FAS included all participants in the APTS who had a valid assessment of the baseline number of weekly attacks and a post-baseline assessment of the number of weekly attacks.
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab
Number analyzed (Participants) | 131
Participants | 17

20. Secondary Outcome: Patient Global Impression of Change (PGIC) Score
Description: The PGIC is a patient-reported measure of improvement in pain sensation and quality of life scored on a scale from 1 (very much improved) to 7 (very much worse). Lower scores indicate better health status.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Eptinezumab
Number analyzed (Participants) | 118
score on a scale
  Week 4: number analyzed (Participants) | 112
  Week 4 | 2.74 (0.12)
  Week 8: number analyzed (Participants) | 95
  Week 8 | 2.69 (0.13)
  Week 12: number analyzed (Participants) | 113
  Week 12 | 2.69 (0.13)
  Week 16: number analyzed (Participants) | 104
  Week 16 | 2.58 (0.13)
  Week 20: number analyzed (Participants) | 91
  Week 20 | 2.72 (0.14)
  Week 24 | 2.58 (0.13)
  Week 28: number analyzed (Participants) | 101
  Week 28 | 2.54 (0.13)
  Week 32: number analyzed (Participants) | 77
  Week 32 | 2.64 (0.13)
  Week 36: number analyzed (Participants) | 111
  Week 36 | 2.58 (0.12)
  Week 40: number analyzed (Participants) | 94
  Week 40 | 2.73 (0.14)
  Week 44: number analyzed (Participants) | 84
  Week 44 | 2.67 (0.13)
  Week 48: number analyzed (Participants) | 96
  Week 48 | 2.65 (0.13)

21. Secondary Outcome: Change From Baseline in Sleep Impact Scale (SIS) Domain Scores Over the Time
Description: The SIS is a patient-reported clinical outcome assessment used to assess quality of life resulting from sleep disturbance. The SIS questionnaire includes 35 items belonging to 7 domains to assess sleep impact on: daily activities; emotional well-being; emotional impact; energy/fatigue; social well-being; mental fatigue; and satisfaction with sleep. Each item, for 6 out of the 7 domains, is rated on a 5-point scale ranging from 1 (always or all of the time) to 5 (never or none of the time), whereas satisfaction with sleep is rated on a 5-point scale ranging from 1 (very satisfied) to 5 (very dissatisfied). Each domain yields a score ranging from 0 to 100, which is presented here. A higher score for Daily Activities, Emotional Well-being, Emotional Impact, Energy/Fatigue, Social Well-being, and Mental Fatigue indicates better quality of life. A lower score for Satisfaction with Sleep indicates a higher quality of life.
Time Frame: Baseline (Week 0), Weeks 4, 12, 16, 24, 28, 36, 40, 48
Population: The FAS included all participants in the APTS who had a valid assessment of the baseline number of weekly attacks and a post-baseline assessment of the number of weekly attacks. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure, and "Number analyzed" is the number of participants evaluable for each specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eptinezumab
Number analyzed (Participants) | 109
score on a scale
  Daily Activities - Week 4: number analyzed (Participants) | 99
  Daily Activities - Week 4 | 14.98 (2.05)
  Daily Activities - Week 12: number analyzed (Participants) | 106
  Daily Activities - Week 12 | 15.26 (2.36)
  Daily Activities - Week 16: number analyzed (Participants) | 92
  Daily Activities - Week 16 | 16.36 (2.48)
  Daily Activities - Week 24 | 15.54 (2.33)
  Daily Activities - Week 28: number analyzed (Participants) | 91
  Daily Activities - Week 28 | 16.17 (2.42)
  Daily Activities - Week 36: number analyzed (Participants) | 99
  Daily Activities - Week 36 | 14.51 (2.39)
  Daily Activities - Week 40: number analyzed (Participants) | 85
  Daily Activities - Week 40 | 17.83 (2.15)
  Daily Activities - Week 48: number analyzed (Participants) | 89
  Daily Activities - Week 48 | 13.29 (2.34)
  Emotional Well-being - Week 4: number analyzed (Participants) | 99
  Emotional Well-being - Week 4 | 17.63 (2.19)
  Emotional Well-being - Week 12: number analyzed (Participants) | 106
  Emotional Well-being - Week 12 | 16.28 (2.32)
  Emotional Well-being - Week 16: number analyzed (Participants) | 92
  Emotional Well-being - Week 16 | 15.72 (2.37)
  Emotional Well-being - Week 24 | 14.04 (2.47)
  Emotional Well-being - Week 28: number analyzed (Participants) | 91
  Emotional Well-being - Week 28 | 17.98 (2.51)
  Emotional Well-being - Week 36: number analyzed (Participants) | 99
  Emotional Well-being - Week 36 | 15.75 (2.34)
  Emotional Well-being - Week 40: number analyzed (Participants) | 85
  Emotional Well-being - Week 40 | 15.40 (2.35)
  Emotional Well-being - Week 48: number analyzed (Participants) | 89
  Emotional Well-being - Week 48 | 14.61 (2.53)
  Emotional Impact - Week 4: number analyzed (Participants) | 99
  Emotional Impact - Week 4 | 17.41 (2.42)
  Emotional Impact - Week 12: number analyzed (Participants) | 106
  Emotional Impact - Week 12 | 17.00 (2.48)
  Emotional Impact - Week 16: number analyzed (Participants) | 92
  Emotional Impact - Week 16 | 18.34 (2.59)
  Emotional Impact - Week 24 | 17.01 (2.42)
  Emotional Impact - Week 28: number analyzed (Participants) | 91
  Emotional Impact - Week 28 | 20.78 (2.53)
  Emotional Impact - Week 36: number analyzed (Participants) | 99
  Emotional Impact - Week 36 | 16.53 (2.53)
  Emotional Impact - Week 40: number analyzed (Participants) | 85
  Emotional Impact - Week 40 | 17.21 (2.57)
  Emotional Impact - Week 48: number analyzed (Participants) | 89
  Emotional Impact - Week 48 | 15.61 (2.58)
  Energy/Fatigue - Week 4: number analyzed (Participants) | 99
  Energy/Fatigue - Week 4 | 16.00 (2.35)
  Energy/Fatigue - Week 12: number analyzed (Participants) | 106
  Energy/Fatigue - Week 12 | 16.67 (2.50)
  Energy/Fatigue - Week 16: number analyzed (Participants) | 92
  Energy/Fatigue - Week 16 | 16.87 (2.63)
  Energy/Fatigue - Week 24 | 16.59 (2.71)
  Energy/Fatigue - Week 28: number analyzed (Participants) | 91
  Energy/Fatigue - Week 28 | 19.67 (2.73)
  Energy/Fatigue - Week 36: number analyzed (Participants) | 99
  Energy/Fatigue - Week 36 | 15.93 (2.62)
  Energy/Fatigue - Week 40: number analyzed (Participants) | 85
  Energy/Fatigue - Week 40 | 19.16 (2.53)
  Energy/Fatigue - Week 48: number analyzed (Participants) | 89
  Energy/Fatigue - Week 48 | 17.65 (2.62)
  Social Well-being - Week 4: number analyzed (Participants) | 99
  Social Well-being - Week 4 | 14.73 (2.06)
  Social Well-being - Week 12: number analyzed (Participants) | 106
  Social Well-being - Week 12 | 15.28 (2.31)
  Social Well-being - Week 16: number analyzed (Participants) | 92
  Social Well-being - Week 16 | 14.68 (2.55)
  Social Well-being - Week 24 | 14.59 (2.46)
  Social Well-being - Week 28: number analyzed (Participants) | 91
  Social Well-being - Week 28 | 17.30 (2.64)
  Social Well-being - Week 36: number analyzed (Participants) | 99
  Social Well-being - Week 36 | 13.27 (2.43)
  Social Well-being - Week 40: number analyzed (Participants) | 85
  Social Well-being - Week 40 | 15.59 (2.42)
  Social Well-being - Week 48: number analyzed (Participants) | 89
  Social Well-being - Week 48 | 14.13 (2.59)
  Mental Fatigue - Week 4: number analyzed (Participants) | 99
  Mental Fatigue - Week 4 | 13.00 (2.23)
  Mental Fatigue - Week 12: number analyzed (Participants) | 106
  Mental Fatigue - Week 12 | 15.00 (2.34)
  Mental Fatigue - Week 16: number analyzed (Participants) | 92
  Mental Fatigue - Week 16 | 15.15 (2.27)
  Mental Fatigue - Week 24 | 13.57 (2.39)
  Mental Fatigue - Week 28: number analyzed (Participants) | 91
  Mental Fatigue - Week 28 | 14.86 (2.36)
  Mental Fatigue - Week 36: number analyzed (Participants) | 99
  Mental Fatigue - Week 36 | 13.64 (2.49)
  Mental Fatigue - Week 40: number analyzed (Participants) | 85
  Mental Fatigue - Week 40 | 13.98 (2.39)
  Mental Fatigue - Week 48: number analyzed (Participants) | 89
  Mental Fatigue - Week 48 | 13.55 (2.42)
  Satisfaction With Sleep - Week 4: number analyzed (Participants) | 99
  Satisfaction With Sleep - Week 4 | -13.86 (2.25)
  Satisfaction With Sleep - Week 12: number analyzed (Participants) | 106
  Satisfaction With Sleep - Week 12 | -13.47 (2.29)
  Satisfaction With Sleep - Week 16: number analyzed (Participants) | 92
  Satisfaction With Sleep - Week 16 | -14.50 (2.40)
  Satisfaction With Sleep - Week 24 | -12.30 (2.20)
  Satisfaction With Sleep - Week 28: number analyzed (Participants) | 91
  Satisfaction With Sleep - Week 28 | -16.67 (2.39)
  Satisfaction With Sleep - Week 36: number analyzed (Participants) | 99
  Satisfaction With Sleep - Week 36 | -13.95 (2.43)
  Satisfaction With Sleep - Week 40: number analyzed (Participants) | 85
  Satisfaction With Sleep - Week 40 | -14.99 (2.60)
  Satisfaction With Sleep - Week 48: number analyzed (Participants) | 89
  Satisfaction With Sleep - Week 48 | -14.19 (2.59)

22. Secondary Outcome: Change From Baseline in EuroQol 5-Dimension 5-Level (EQ-5D-5L) Score at Weeks 4, 16, 28, 40 and 48
Description: The EQ-5D-5L is a patient-reported assessment designed to measure the participant's well-being. It consists of 5 descriptive items (mobility, self-care, usual activities, pain/discomfort, and depression/anxiety). Each descriptive item is rated on a 5-point index ranging from 1 (no problems) to 5 (extreme problems).
Time Frame: Baseline (Week 0), Weeks 4, 16, 28, 40, 48
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eptinezumab
Number analyzed (Participants) | 97
score on a scale
  Mobility - Week 4 | 0.1 (0.89)
  Self Care - Week 4 | 0.0 (0.47)
  Usual Activities - Week 4 | -0.2 (1.13)
  Pain/Discomfort - Week 4 | -0.1 (1.28)
  Anxiety/Depression - Week 4 | -0.1 (0.70)
  Mobility - Week 16: number analyzed (Participants) | 90
  Mobility - Week 16 | 0.1 (1.02)
  Self Care - Week 16: number analyzed (Participants) | 90
  Self Care - Week 16 | 0.0 (0.69)
  Usual Activities - Week 16: number analyzed (Participants) | 90
  Usual Activities - Week 16 | -0.2 (1.07)
  Pain/Discomfort - Week 16: number analyzed (Participants) | 90
  Pain/Discomfort - Week 16 | -0.2 (1.48)
  Anxiety/Depression - Week 16: number analyzed (Participants) | 90
  Anxiety/Depression - Week 16 | -0.1 (0.98)
  Mobility - Week 28: number analyzed (Participants) | 89
  Mobility - Week 28 | 0.1 (0.92)
  Self Care - Week 28: number analyzed (Participants) | 89
  Self Care - Week 28 | 0.1 (0.65)
  Usual Activities - Week 28: number analyzed (Participants) | 89
  Usual Activities - Week 28 | -0.1 (1.14)
  Pain/Discomfort - Week 28: number analyzed (Participants) | 89
  Pain/Discomfort - Week 28 | -0.1 (1.26)
  Anxiety/Depression - Week 28: number analyzed (Participants) | 89
  Anxiety/Depression - Week 28 | -0.1 (0.98)
  Mobility - Week 40: number analyzed (Participants) | 83
  Mobility - Week 40 | 0.0 (0.96)
  Self Care - Week 40: number analyzed (Participants) | 83
  Self Care - Week 40 | 0.0 (0.49)
  Usual Activities - Week 40: number analyzed (Participants) | 83
  Usual Activities - Week 40 | -0.4 (1.04)
  Pain/Discomfort - Week 40: number analyzed (Participants) | 83
  Pain/Discomfort - Week 40 | -0.3 (1.42)
  Anxiety/Depression - Week 40: number analyzed (Participants) | 83
  Anxiety/Depression - Week 40 | -0.1 (0.97)
  Mobility - Week 48: number analyzed (Participants) | 85
  Mobility - Week 48 | -0.0 (0.90)
  Self Care - Week 48: number analyzed (Participants) | 85
  Self Care - Week 48 | 0.0 (0.53)
  Usual Activities - Week 48: number analyzed (Participants) | 85
  Usual Activities - Week 48 | -0.2 (1.17)
  Pain/Discomfort - Week 48: number analyzed (Participants) | 85
  Pain/Discomfort - Week 48 | -0.1 (1.24)
  Anxiety/Depression - Week 48: number analyzed (Participants) | 85
  Anxiety/Depression - Week 48 | -0.0 (1.04)

23. Secondary Outcome: Change From Baseline in the EQ-5D-5L Visual Analog Scale (VAS) Score at Weeks 4, 16, 28, 40 and 48
Description: The EQ-5D-5L VAS is a participant-reported assessment designed to measure the participant's well-being and ranges from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline (Week 0), Weeks 4, 16, 28, 40, 48
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Eptinezumab
Number analyzed (Participants) | 97
score on a scale
  Week 4 | 9.03 (2.07)
  Week 16: number analyzed (Participants) | 90
  Week 16 | 9.26 (2.30)
  Week 28: number analyzed (Participants) | 89
  Week 28 | 6.99 (2.39)
  Week 40: number analyzed (Participants) | 83
  Week 40 | 8.61 (2.11)
  Week 48: number analyzed (Participants) | 85
  Week 48 | 6.90 (2.31)

24. Secondary Outcome: Change From Baseline in the Work Productivity Activity Impairment: General Health Second Version (WPAI:GH2.0) Sub-Scores (Absenteeism, Presenteeism, Work Productivity Loss, Activity Impairment) at Weeks 4, 16, 28, 40 and 48
Description: The WPAI:GH2.0 is a patient self-rated clinical outcome assessment designed to provide a quantitative measure of the work productivity and activity impairment due to a health condition. The WPAI:GH2.0 assesses activities over the preceding 7 days and consists of 6 items: 1 item assesses employment (yes/no); 3 items assess the number of hours worked, the number of hours missed from work due to the participant's condition, or due to other reasons; and 2 visual numerical scales assess how much the participant's condition affects his/her productivity at work and his/her ability to complete normal daily activities. Each item (Absenteeism, Presenteeism, Work Productivity Loss, Activity Impairment) was calculated into an impairment percentage ranging from 0 to 100%, with higher numbers indicating greater impairment and less productivity (i.e. worse outcomes). Change from baseline for each item is shown here.
Time Frame: Baseline (Week 0), Weeks 4, 16, 28, 40, 48
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eptinezumab
Number analyzed (Participants) | 95
score on a scale
  Absenteeism - Week 4: number analyzed (Participants) | 50
  Absenteeism - Week 4 | -12.03 (2.82)
  Absenteeism - Week 16: number analyzed (Participants) | 44
  Absenteeism - Week 16 | -8.19 (2.98)
  Absenteeism - Week 28: number analyzed (Participants) | 42
  Absenteeism - Week 28 | -12.73 (1.70)
  Absenteeism - Week 40: number analyzed (Participants) | 39
  Absenteeism - Week 40 | -12.05 (2.29)
  Absenteeism - Week 48: number analyzed (Participants) | 46
  Absenteeism - Week 48 | -5.30 (2.99)
  Presenteeism - Week 4: number analyzed (Participants) | 45
  Presenteeism - Week 4 | -14.29 (3.23)
  Presenteeism - Week 16: number analyzed (Participants) | 39
  Presenteeism - Week 16 | -14.54 (3.74)
  Presenteeism - Week 28: number analyzed (Participants) | 38
  Presenteeism - Week 28 | -11.86 (3.78)
  Presenteeism - Week 40: number analyzed (Participants) | 35
  Presenteeism - Week 40 | -9.88 (3.58)
  Presenteeism - Week 48: number analyzed (Participants) | 41
  Presenteeism - Week 48 | -12.70 (3.53)
  Work productivity loss - Week 4: number analyzed (Participants) | 45
  Work productivity loss - Week 4 | -17.28 (3.34)
  Work productivity loss - Week 16: number analyzed (Participants) | 39
  Work productivity loss - Week 16 | -16.53 (3.98)
  Work productivity loss - Week 28: number analyzed (Participants) | 38
  Work productivity loss - Week 28 | -14.60 (3.96)
  Work productivity loss - Week 40: number analyzed (Participants) | 35
  Work productivity loss - Week 40 | -12.50 (3.78)
  Work productivity loss - Week 48: number analyzed (Participants) | 41
  Work productivity loss - Week 48 | -12.16 (3.77)
  Activity impairment - Week 4 | -15.99 (2.56)
  Activity impairment - Week 16: number analyzed (Participants) | 89
  Activity impairment - Week 16 | -15.64 (2.84)
  Activity impairment - Week 28: number analyzed (Participants) | 88
  Activity impairment - Week 28 | -17.37 (2.74)
  Activity impairment - Week 40: number analyzed (Participants) | 82
  Activity impairment - Week 40 | -18.73 (2.79)
  Activity impairment - Week 48: number analyzed (Participants) | 84
  Activity impairment - Week 48 | -14.35 (2.95)

25. Secondary Outcome: Health Care Resource Utilization - Number of Visits to a Family Doctor/General Practitioner
Description: Number of participants who visited a family doctor/general practitioner has been reported.
Time Frame: Baseline (Week 0), Weeks 4, 16, 28, 40, 48
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab
Number analyzed (Participants) | 112
Participants
  Week 0 - 0 visits | 81
  Week 0 - 1 visit | 18
  Week 0 - 2 visits | 10
  Week 0 - 3 visits | 1
  Week 0 - 4 visits | 2
  Week 4 - 0 visits: number analyzed (Participants) | 105
  Week 4 - 0 visits | 82
  Week 4 - 1 visit: number analyzed (Participants) | 105
  Week 4 - 1 visit | 17
  Week 4 - 2 visits: number analyzed (Participants) | 105
  Week 4 - 2 visits | 5
  Week 4 - 3 visits: number analyzed (Participants) | 105
  Week 4 - 3 visits | 1
  Week 16 - 0 visits: number analyzed (Participants) | 101
  Week 16 - 0 visits | 80
  Week 16 - 1 visit: number analyzed (Participants) | 101
  Week 16 - 1 visit | 15
  Week 16 - 2 visits: number analyzed (Participants) | 101
  Week 16 - 2 visits | 2
  Week 16 - 3 visits: number analyzed (Participants) | 101
  Week 16 - 3 visits | 2
  Week 16 - 4 visits: number analyzed (Participants) | 101
  Week 16 - 4 visits | 1
  Week 16 - 5 visits: number analyzed (Participants) | 101
  Week 16 - 5 visits | 1
  Week 28 - 0 visits: number analyzed (Participants) | 100
  Week 28 - 0 visits | 76
  Week 28 - 1 visit: number analyzed (Participants) | 100
  Week 28 - 1 visit | 14
  Week 28 - 2 visits: number analyzed (Participants) | 100
  Week 28 - 2 visits | 6
  Week 28 - 3 visits: number analyzed (Participants) | 100
  Week 28 - 3 visits | 4
  Week 40 - 0 visits: number analyzed (Participants) | 91
  Week 40 - 0 visits | 67
  Week 40 - 1 visit: number analyzed (Participants) | 91
  Week 40 - 1 visit | 13
  Week 40 - 2 visits: number analyzed (Participants) | 91
  Week 40 - 2 visits | 8
  Week 40 - 3 visits: number analyzed (Participants) | 91
  Week 40 - 3 visits | 1
  Week 40 - 6 visits: number analyzed (Participants) | 91
  Week 40 - 6 visits | 2
  Week 48 - 0 visits: number analyzed (Participants) | 94
  Week 48 - 0 visits | 78
  Week 48 - 1 visit: number analyzed (Participants) | 94
  Week 48 - 1 visit | 9
  Week 48 - 2 visits: number analyzed (Participants) | 94
  Week 48 - 2 visits | 5
  Week 48 - 3 visits: number analyzed (Participants) | 94
  Week 48 - 3 visits | 1
  Week 48 - 6 visits: number analyzed (Participants) | 94
  Week 48 - 6 visits | 1

26. Secondary Outcome: Health Care Resource Utilization - Number of Visits to a Specialist
Description: Number of participants who visited a specialist has been reported.
Time Frame: Baseline (Week 0), Weeks 4, 16, 28, 40, 48
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab
Number analyzed (Participants) | 112
Participants
  Week 0 - 0 visits | 51
  Week 0 - 1 visit | 40
  Week 0 - 2 visits | 18
  Week 0 - 3 visits | 2
  Week 0 - 6 visits | 1
  Week 4 - 0 visits: number analyzed (Participants) | 105
  Week 4 - 0 visits | 74
  Week 4 - 1 visit: number analyzed (Participants) | 105
  Week 4 - 1 visit | 28
  Week 4 - 2 visits: number analyzed (Participants) | 105
  Week 4 - 2 visits | 1
  Week 4 - 3 visits: number analyzed (Participants) | 105
  Week 4 - 3 visits | 1
  Week 4 - 4 visits: number analyzed (Participants) | 105
  Week 4 - 4 visits | 1
  Week 16 - 0 visits: number analyzed (Participants) | 101
  Week 16 - 0 visits | 64
  Week 16 - 1 visit: number analyzed (Participants) | 101
  Week 16 - 1 visit | 23
  Week 16 - 2 visits: number analyzed (Participants) | 101
  Week 16 - 2 visits | 9
  Week 16 - 3 visits: number analyzed (Participants) | 101
  Week 16 - 3 visits | 2
  Week 16 - 4 visits: number analyzed (Participants) | 101
  Week 16 - 4 visits | 1
  Week 16 - 5 visits: number analyzed (Participants) | 101
  Week 16 - 5 visits | 1
  Week 16 - 7 visits: number analyzed (Participants) | 101
  Week 16 - 7 visits | 1
  Week 28 - 0 visits: number analyzed (Participants) | 100
  Week 28 - 0 visits | 68
  Week 28 - 1 visit: number analyzed (Participants) | 100
  Week 28 - 1 visit | 25
  Week 28 - 2 visits: number analyzed (Participants) | 100
  Week 28 - 2 visits | 4
  Week 28 - 4 visits: number analyzed (Participants) | 100
  Week 28 - 4 visits | 2
  Week 28 - 5 visits: number analyzed (Participants) | 100
  Week 28 - 5 visits | 1
  Week 40 - 0 visits: number analyzed (Participants) | 91
  Week 40 - 0 visits | 62
  Week 40 - 1 visit: number analyzed (Participants) | 91
  Week 40 - 1 visit | 22
  Week 40 - 2 visits: number analyzed (Participants) | 91
  Week 40 - 2 visits | 4
  Week 40 - 3 visits: number analyzed (Participants) | 91
  Week 40 - 3 visits | 1
  Week 40 - 4 visits: number analyzed (Participants) | 91
  Week 40 - 4 visits | 1
  Week 40 - 6 visits: number analyzed (Participants) | 91
  Week 40 - 6 visits | 1
  Week 48 - 0 visits: number analyzed (Participants) | 94
  Week 48 - 0 visits | 72
  Week 48 - 1 visit: number analyzed (Participants) | 94
  Week 48 - 1 visit | 17
  Week 48 - 2 visits: number analyzed (Participants) | 94
  Week 48 - 2 visits | 3
  Week 48 - 3 visits: number analyzed (Participants) | 94
  Week 48 - 3 visits | 1
  Week 48 - 6 visits: number analyzed (Participants) | 94
  Week 48 - 6 visits | 1

27. Secondary Outcome: Health Care Resource Utilization - Number of Emergency Department Visits Due to Cluster Headache
Description: Number of participants who visited an emergency department due to CH has been reported.
Time Frame: Baseline (Week 0), Weeks 4, 16, 28, 40, 48
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab
Number analyzed (Participants) | 112
Participants
  Week 0 - 0 visits | 108
  Week 0 - 1 visit | 1
  Week 0 - 2 visits | 1
  Week 0 - 4 visits | 2
  Week 4 - 0 visits: number analyzed (Participants) | 105
  Week 4 - 0 visits | 102
  Week 4 - 1 visit: number analyzed (Participants) | 105
  Week 4 - 1 visit | 2
  Week 4 - 4 visits: number analyzed (Participants) | 105
  Week 4 - 4 visits | 1
  Week 16 - 0 visits: number analyzed (Participants) | 101
  Week 16 - 0 visits | 97
  Week 16 - 1 visit: number analyzed (Participants) | 101
  Week 16 - 1 visit | 2
  Week 16 - 2 visits: number analyzed (Participants) | 101
  Week 16 - 2 visits | 1
  Week 16 - 4 visits: number analyzed (Participants) | 101
  Week 16 - 4 visits | 1
  Week 28 - 0 visits: number analyzed (Participants) | 100
  Week 28 - 0 visits | 96
  Week 28 - 1 visit: number analyzed (Participants) | 100
  Week 28 - 1 visit | 2
  Week 28 - 2 visits: number analyzed (Participants) | 100
  Week 28 - 2 visits | 1
  Week 28 - 4 visits: number analyzed (Participants) | 100
  Week 28 - 4 visits | 1
  Week 40 - 0 visits: number analyzed (Participants) | 91
  Week 40 - 0 visits | 88
  Week 40 - 1 visit: number analyzed (Participants) | 91
  Week 40 - 1 visit | 1
  Week 40 - 2 visits: number analyzed (Participants) | 91
  Week 40 - 2 visits | 2
  Week 48 - 0 visits: number analyzed (Participants) | 94
  Week 48 - 0 visits | 91
  Week 48 - 1 visit: number analyzed (Participants) | 94
  Week 48 - 1 visit | 1
  Week 48 - 2 visits: number analyzed (Participants) | 94
  Week 48 - 2 visits | 1
  Week 48 - 3 visits: number analyzed (Participants) | 94
  Week 48 - 3 visits | 1

28. Secondary Outcome: Health Care Resource Utilization - Number of Hospital Admissions Due to Cluster Headache
Description: Number of participants admitted to the hospital due to CH has been reported.
Time Frame: Baseline (Week 0), Weeks 4, 16, 28, 40, 48
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab
Number analyzed (Participants) | 112
Participants
  Week 0 - 0 admissions | 110
  Week 0 - 1 admission | 2
  Week 4 - 0 admissions: number analyzed (Participants) | 105
  Week 4 - 0 admissions | 103
  Week 4 - 1 admission: number analyzed (Participants) | 105
  Week 4 - 1 admission | 2
  Week 16 - 0 admissions: number analyzed (Participants) | 101
  Week 16 - 0 admissions | 98
  Week 16 - 1 admission: number analyzed (Participants) | 101
  Week 16 - 1 admission | 2
  Week 16 - 5 admissions: number analyzed (Participants) | 101
  Week 16 - 5 admissions | 1
  Week 28 - 0 admissions: number analyzed (Participants) | 100
  Week 28 - 0 admissions | 97
  Week 28 - 1 admission: number analyzed (Participants) | 100
  Week 28 - 1 admission | 3
  Week 40 - 0 admissions: number analyzed (Participants) | 91
  Week 40 - 0 admissions | 89
  Week 40 - 1 admission: number analyzed (Participants) | 91
  Week 40 - 1 admission | 1
  Week 40 - 5 admissions: number analyzed (Participants) | 91
  Week 40 - 5 admissions | 1
  Week 48 - 0 admissions: number analyzed (Participants) | 94
  Week 48 - 0 admissions | 92
  Week 48 - 1 admission: number analyzed (Participants) | 94
  Week 48 - 1 admission | 2

29. Secondary Outcome: Health Care Resource Utilization - Total Number of Overnight Hospital Stays Due to Cluster Headache
Description: Number of participants who had overnight hospital stays due to CH has been reported.
Time Frame: Baseline (Week 0), Weeks 4, 16, 28, 40, 48
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab
Number analyzed (Participants) | 112
Participants
  Week 0 - 0 visits | 109
  Week 0 - 1 visit | 2
  Week 0 - 2 visits | 1
  Week 4 - 0 visits: number analyzed (Participants) | 105
  Week 4 - 0 visits | 105
  Week 16 - 0 visits: number analyzed (Participants) | 101
  Week 16 - 0 visits | 98
  Week 16 - 1 visit: number analyzed (Participants) | 101
  Week 16 - 1 visit | 1
  Week 16 - 7 visits: number analyzed (Participants) | 101
  Week 16 - 7 visits | 1
  Week 16 - 10 visits: number analyzed (Participants) | 101
  Week 16 - 10 visits | 1
  Week 28 - 0 visits: number analyzed (Participants) | 100
  Week 28 - 0 visits | 99
  Week 28 - 1 visit: number analyzed (Participants) | 100
  Week 28 - 1 visit | 1
  Week 40 - 0 visits: number analyzed (Participants) | 91
  Week 40 - 0 visits | 90
  Week 40 - 1 visit: number analyzed (Participants) | 91
  Week 40 - 1 visit | 1
  Week 48 - 0 visits: number analyzed (Participants) | 94
  Week 48 - 0 visits | 92
  Week 48 - 1 visit: number analyzed (Participants) | 94
  Week 48 - 1 visit | 1
  Week 48 - 5 visits: number analyzed (Participants) | 94
  Week 48 - 5 visits | 1

ADVERSE EVENTS:
Time Frame: From the day of first dose of study drug (Baseline [Week 0]) up to Week 56
Description: The APTS included all participants who received infusion with eptinezumab
Arm/Group | Eptinezumab
All-Cause Mortality (participants affected / at risk) | 0/131
Serious Adverse Events (participants affected / at risk) | 11/131
Other Adverse Events (participants affected / at risk) | 96/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eptinezumab (N=131)
Thyroiditis acute (Endocrine disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cluster headache (Nervous system disorders) | 1 (7)
Suicide attempt (Psychiatric disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eptinezumab (N=131)
Atrioventricular block first degree (Cardiac disorders) | 3 (5)
Tinnitus (Ear and labyrinth disorders) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 4 (6)
Constipation (Gastrointestinal disorders) | 6 (9)
Nausea (Gastrointestinal disorders) | 8 (8)
Vomiting (Gastrointestinal disorders) | 7 (7)
Asthenia (General disorders) | 6 (11)
Fatigue (General disorders) | 22 (30)
Influenza like illness (General disorders) | 3 (4)
Oedema peripheral (General disorders) | 5 (7)
Bronchitis (Infections and infestations) | 3 (3)
COVID-19 (Infections and infestations) | 29 (31)
Gastroenteritis (Infections and infestations) | 3 (3)
Influenza (Infections and infestations) | 10 (10)
Nasopharyngitis (Infections and infestations) | 24 (33)
Pharyngitis (Infections and infestations) | 5 (5)
Pneumonia (Infections and infestations) | 3 (4)
Rhinitis (Infections and infestations) | 6 (6)
Sinusitis (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 4 (5)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 3 (4)
Blood triglycerides increased (Investigations) | 3 (3)
Weight increased (Investigations) | 8 (8)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Dizziness (Nervous system disorders) | 7 (7)
Insomnia (Psychiatric disorders) | 8 (9)
Nightmare (Psychiatric disorders) | 3 (3)
Sleep disorder (Psychiatric disorders) | 3 (3)
Suicidal ideation (Psychiatric disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9)
Hypertension (Vascular disorders) | 4 (4)
Orthostatic hypotension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/97/NCT05064397/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT05064397/SAP_002.pdf